CLINICAL TRIAL: NCT07200232
Title: Clinical Assessment of ECG Signal Quality With the ZywieZ3 Sensor and Adhesive Versus a Traditional Device Over a 1 Hour Period, Monitoring Skin Adhesion / ECG Performance of the ZywieZ3 Sensor and Adhesive Over 10 Days, and of the Effects of Variable ECG Electrode Placement With the ZywieZ3 Sensor and Adhesive
Brief Title: A Three-phase Study That Will Compare the ECG Data Recorded Using the Test Device With the Data Recorded by a Reference Device, Evaluate the ECG Signal Quality of the Test Device Over a 10-day Simulated Use Period, and Assess the Effects of Variable ECG Electrode Placement for the Test Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zywie, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2410001-150
Record Dates: First submitted 2025-09-12; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Healthy Subjects
Keywords: ECG Signal Quality Evaluation; Variable ECG Electrode Placement; Skin Adhesion of ECG Device and Adhesive; ECG Device and Adhesive versus Traditional ECG Device

STUDY DESIGN:
Intervention Model Description: For Phase 1 and Phase 2, a single group of at least 25 subjects will participate in both study phases, wearing a test and reference device for 1 hour and then the test device for a 10-day test period. For Phase 3, a single group of at least 20 subjects will participate in this study for a single test day with 15-minute ECG readings performed with the test device at the ideal location (control) and again with the test device applied to the skin in nine incorrect test locations/orientations (test positions).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Phase 1 Test Device Application and comparison to Reference Device (Other): Subjects apply Test Device Sensor and Adhesive according to instructions. Analysts apply Reference Device. Subject wears both devices for 1-hour with ECG Readings collected and compared between the two devices.
  Interventions: Device: Phase 1 Test Device Sensor and Adhesive and Reference Device
- Phase 2 Test Device Sensor and Adhesive (Other): Test Device Sensor and Adhesive consisting of a single sensor applied to an adhesive than is then applied to the upper-left chest area of a subject for 10 days
  Interventions: Device: Phase 2 Test Device ECG Signal quality over a 10-day simulated use period
- Phase 3 Variable placement of the Test Device Sensor and Adhesive (Other): Assess the effects of variable ECG electrode placement for the Test Device Sensor and Adhesive for producing relevant ECG data
  Interventions: Device: Test Device Sensor and Adhesive Variable Placement

INTERVENTIONS:
Device: Phase 1 Test Device Sensor and Adhesive and Reference Device — Test Device Sensor and Adhesive and Reference Device ECG Data Collection for 1 hour
  Arms: Phase 1 Test Device Application and comparison to Reference Device
Device: Phase 2 Test Device ECG Signal quality over a 10-day simulated use period — Evaluation of the ECG-signal quality of the Test Device sensor and adhesive applied to a single site on a subject's chest to collect ECG readings for a 10-day period.
  Arms: Phase 2 Test Device Sensor and Adhesive
Device: Test Device Sensor and Adhesive Variable Placement — Comparison of nine incorrect locations of Test Device Sensor and Adhesive to the ideal location
  Arms: Phase 3 Variable placement of the Test Device Sensor and Adhesive

SUMMARY:
This clinical study will be performed in three phases.

The purpose of Phase 1 of this study is to compare the ECG data recorded using the ZywieZ3 Sensor and ZywieZ3 Adhesive ("Test Device") to the data recorded by a traditional 3-lead ECG device that uses wet Ag-AgCl adhesives in a standard lead location ("Reference Device"). The ECG signals will be recorded simultaneously with both ECG devices from the subjects in conditions that represent the devices' intended use for 1 hour. This comparison will determine whether the Test Device recordings are similar to the "gold standard" Reference Device. The testing methodology for this portion of the study is based on guidance provided by the FDA to the Sponsor.

The purpose of Phase 2 of this study is to evaluate the ECG signal quality of the Test Device over a 10-day simulated use period by human subjects. This duration of 10 days represents the expected maximum period of usage for the Test Device by the Sponsor. The skin adhesion properties of the Test Device will be evaluated, including a determination of whether any skin reactions, discoloration of the Test Device adhesive (including the snaps and hydrogel), or Test Device adhesive degradation leading to particulate formation occurs over a 10-day simulated use period by human subjects. During this testing, a human factor critical task analysis will be conducted via a collection of observational data regarding success in subject completion of Sponsor-identified critical tasks, subject completion of knowledge questionnaires relating to aspects of Sponsor-identified critical tasks, and subject completion of general subjective questionnaires regarding any difficulty they experienced with use of the Test Device. Testing methodology for this portion of the study is based upon the "Adhesive Performance (Duration of Use)" [Section 5.4] procedures from ANSI/AAMI Standard EC12:2000/(R)2020, Disposable ECG Electrodes and the 2016 FDA Guidance for Industry and Food and Drug Administration Staff titled "Applying Human Factors and Usability Engineering to Medical Devices."

The purpose of Phase 3 of this clinical study is to assess the effects of variable ECG electrode placement for the ZywieZ3 Sensor and ZywieZ3 Adhesive ("Test Device"). This testing is intended to determine whether ECG electrode placement variability produces unacceptable / non-clinically relevant ECG data and what level of ECG electrode placement variability is acceptable.

DETAILED DESCRIPTION:
For Phase 1 and Phase 2, at least 25 subjects will participate in both study phases wearing a test and reference device for 1 hour and then the test device for a 10-day test period. Subjects will apply the Test Device on their skin by following the Sponsor-provided instructions. A Testing Facility analyst will conduct an initial visual evaluation of the level of skin adhesion for the Test Device and then apply the Reference Device to the subjects' chest. ECG data collection will be initiated for the Test Device and Reference Device by subjects and a Testing Facility analyst, respectively. During ECG data collection initiation, a Testing Facility analyst, following the 2016 FDA Guidance for Industry and Food and Drug Administration Staff titled "Applying Human Factors and Usability Engineering to Medical Devices," will collect observational data regarding each subject's success or failure to complete Sponsor-identified critical tasks correctly. Following ECG data collection initiation, subjects will complete a knowledge questionnaire to determine whether they fully understood Sponsor-identified critical tasks and a general subjective questionnaire regarding any difficulty they experienced with the use of the Test Device. Subjects will observe a 5-minute stabilization period to ensure that both devices are connected appropriately and have a stable input signal. Following the stabilization period, 25 minutes of ECG data will be collected while subjects are sitting idle. Subjects will then complete three standardized 10-minute activity periods of standing up, lying down, and repeatedly transitioning from lying down to standing up while ECG data are collected by the Test Device and Reference Device, completing a 60-minute data collection. After completing the 1-hour ECG data collection period, the reference device will be removed. Approximately 1 hour after the removal of the Reference Device, a trained Testing Facility analyst will visually score the skin condition at the relevant reference adhesive application sites. The subjects will be allowed to leave the Testing Facility and continue wearing the Test Device for 10 days. Subjects will be instructed to follow the Sponsor-provided instructions for use during this time period.

For Phase 1, subjects will be shown an instructional video and read the patient guide included in the sensor kit. Subjects will then be asked to apply the Test device themselves. A Testing Facility analyst will collect observational data regarding each subject's success or failure to complete Sponsor-identified critical tasks correctly, and the subject will complete a knowledge questionnaire to determine whether they fully understood Sponsor-identified critical tasks. The Testing Facility analyst will measure the Test device placement offset after subjects have applied the device to themselves. If the device is placed grossly incorrectly, the Training Facility Analyst will note the issue and guide the subject in correcting the adhesive placement. The analyst will not physically adjust the placement but will only provide guidance, similar to how Zywie's customer support would guide over the phone when incorrect data is identified during production use. The Sponsor will download ECG data from the Test Device from the initial 1-hour ECG data collection period from cloud-based data repositories. The testing facility will provide the Reference Device data to the Sponsor for data analysis according to the statistical analysis plan. The analysis results will be included as an appendix to the study's final report upon completion. Two cardiologists contracted by the Sponsor will independently review de-identified ECG data recorded using both devices in accordance with the statistical analysis plan. A third cardiologist, also contracted by the Sponsor, will be employed to review the ECG data collected if the first two do not agree with their assessment.

For Phase 2 on Day 10, subjects will return to the Testing Facility for a final visual evaluation of the level of skin adhesion of the Test Device by a trained Testing Facility analyst. The subject will then remove the Test Device, and a trained Testing Facility analyst will visually examine the Test Device Adhesive for any discoloration (including snaps and hydrogel) or particulate formation. At 1 hour after removal of the Test Device, a trained Testing Facility analyst will visually evaluate the skin condition at the adhesive application site.

For Phase 2, the Sponsor will download ECG data for the Test Device following the 10-day period from a cloud-based data repository for data analysis according to the statistical analysis plan. Two cardiologists contracted by the Sponsor will review the collected ECG data to determine whether the Test Device produced clinically relevant ECG data during the entire 10-day wear time. A third cardiologist, also contracted by the Sponsor, will be employed to review the ECG data collected if the first two do not agree with their assessment. Upon completion of the analysis, the analysis results will be appended to the study's final report. Skin adhesion scores and skin condition evaluations will also be summarized, and the Testing Facility will conduct a descriptive statistical analysis for each visual evaluation time point. Summaries of electrode discoloration/particulate observation evaluations will also be prepared.

For Phase 3, at least 20 subjects will participate in this study for a single test day. A testing facility analyst will apply the test device to the ideal location (control). The subjects will wear the Test Device for 15 minutes of ECG recording. The test device will then be applied to the skin in nine incorrect test locations/orientations (test positions) for all subjects as described in Appendix 2, Table 5, and worn for an additional 15 minutes of ECG recording for each test position. A statistical analysis of ECG recordings from the electrode placements will be conducted. Two cardiologists contracted by the Sponsor will independently review the ECG data recorded for the Test Device applied to the ideal (control) and 9 incorrect test locations/orientations in accordance with the statistical analysis plan. A third cardiologist, also contracted by the Sponsor, will be employed to review the ECG data collected if the first two do not agree with their assessment. Upon completion of the analysis, the analysis results will be appended to the study's final report.

ELIGIBILITY:
Inclusion Criteria:

* Of the 25 subjects for Phase 1 and 2 and 20 subjects for Phase 3 who complete the study, at least 40% of subjects must be male, and at least 40% of the subjects must be female.
* Of the 25 subjects for Phase 1 and 2 and 20 subjects for Phase 3 who complete the study, no more than 50% may be white/Caucasian, and at least 50% must be classified as each of the following races: Asian, Black / African American, American Indian / Alaskan Native, and Native Hawaiian / Pacific Islander.
* Subjects must be 21 to 80 years of age. Of the 25 subjects for Phase 1 and 2 and 20 subjects for Phase 3 who complete the study, no more than 30% can be from a given quartile (21 to 36, 36 to 51, 51 to 65, and 65 to 80 year of age) of the age range.
* Subjects' body mass index (BMI) will be calculated based on their weight and height at the time of consent. BMI will be calculated using the CDC's online Adult BMI Calculator. This calculator will also automatically categorize the calculated BMI as underweight (< 18.5), healthy (18.5 to 24.9), overweight (25.0 to 29.9), or obese (≥ 30.0). Of the 25 subjects for Phase 1 and 2 and 20 subjects for Phase 3 who complete the study, no more than 30% can be from a given BMI category.
* Subjects' education will be categorized as high school / GED, associate college degree, bachelor college degree, or post-graduate degree (e.g., M.S. or Ph.D.). Of the 25 subjects who complete Phases 1 and 2 of the study, no more than 7 subjects can be from a given educational level category.
* Of the 25 subjects who complete Phases 1 and 2 of the study, at least 7 must self-report some type of limited hand/arm dexterity.
* Subjects must be able to read, write, and understand English.
* Subjects must be in good general health (i.e., no current or recent severe illness).
* All subjects with body hair on their upper-left chest must be willing to have the body hair clipped by a Testing Facility analyst before application of the Test Device.
* Subjects participating in Phase 1 must be willing to have the body hair clipped by a Testing Facility analyst from the right clavicular region and middle of their left rib cage.
* Subjects participating in Phases 1 and 2 must be willing to clean the skin of the right clavicular region, upper-left chest, and middle of their left rib cage with 70% isopropanol preparation pads prior to their application of the Test Device and application of the Reference Device by a Testing Facility analyst. Subjects participating in Phase 3 must be willing to clean the skin of the upper-left chest with 70% isopropanol preparation pads before application of the Test Device.

Exclusion Criteria:

* Subjects cannot be currently participating in another clinical study.
* Subjects cannot have active skin rashes, dermatoses, or breaks in the skin on their clavicles, and the middle of their left rib cage for Phase 1 and 2 or on the upper left chest region for all phases.
* Subjects cannot have undergone any surgeries during the last 3 months involving incisions along their clavicles and the middle of their left rib cage for Phase 1 and Phase 2 or on the upper left chest region for all phases.
* Subjects cannot have any tattoos on their clavicles and the middle of their left rib cage for Phase 1 and Phase 2 or on the upper left chest region for all phases.
* Subjects cannot have currently inflammatory skin conditions (e.g., atopic dermatitis/eczema, contact dermatitis, or psoriasis) anywhere on the body within 2 days of the start of the test period and during the test period.
* Subjects cannot have a medical diagnosis of an organ transplant, medicated or uncontrolled diabetes, hepatitis B, hepatitis C, an immunocompromised condition such as AIDS (or HIV positive), lupus, medicated fibromyalgia, ulcerative colitis, Crohn's disease, moderate to severe asthma (requiring daily use of medication), or medicated multiple sclerosis.
* Subjects cannot have a pacemaker.
* Subjects cannot have any type of port, shunt, or Peripherally Inserted Central Catheter (PICC).
* Subjects cannot receive any vaccinations within 7 days of the start of the test period and while participating in the single-day or 10-day test period.
* Subjects cannot have known allergies or sensitivities to latex (natural rubber), adhesives, inks, sunscreens, deodorants, laundry detergents, cleansers, soaps, lotions, to topical application of fragrances (e.g., perfumes or colognes), acrylic, hydrogel, isopropyl alcohol, C11-12 isoparaffin, isopropyl palmitate, isopropyl myristate, or isopropyl stearate.
* Subjects participating in Phases 1 and 2 cannot use antihistamines within 2 days of the start of the test period through to the completion of the 10-day test period, which may interfere with the evaluation of skin reactions after application of the devices.
* Subjects cannot be pregnant or plan to become pregnant / impregnate a sexual partner during the study.
* Subjects cannot be nursing a child during the study.
* Subjects cannot have any medical condition or use any medications that, in the opinion of the Principal Investigator or Consulting Physicians, should preclude participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Phase 1: Test Device Sensor and Adhesive Equivalence to a Reference Device | From enrollment to end of the 1-hour ECG reading period
  ECG recordings will be simultaneously collected from 25 subjects using the test and reference devices for one hour, during which subjects will perform a controlled activity for 55 minutes, including sitting, standing, and lying down. The clinical ECG interpretation will be performed independently by two board-certified cardiologists, with a third involved when there is a disagreement between the two. Two full-disclosure reports with de-identified ECG strips and timestamp information, one for each Test and Reference device, will be shared with the cardiologists. Each cardiologist will review reports and assess the overall quality of the ECG waveform, focusing on amplitude and morphology. The cardiologists will provide their assessment as 'Interpretable' with normal sinus rhythm, ectopy [≤ 3 consecutive beats], or any arrhythmia, or 'Uninterpretable' as noisy or not readable data. For each 3-minute ECG segment, a conclusion of 'equivalent or better' will be based on the assessments.
Phase 2: Evaluate the ECG signal quality of the Test Device over a 10-day simulated use period by human subjects | From enrollment to 10 days after initial application of the Test Device
  ECG recordings will be collected from 25 subjects using the ZywieZ3 device over 10 days. During this period, subjects will perform routine activities. For each subject, a report with ECG recordings from 10 days duration will be created. Each cardiologist will review the ECG data recorded and assess the clinical interpretability of the ECG waveform. Cardiologist will assess a page of data from every 12-hour window (consisting of 30 minutes of data) and stop if at least a 30-second ECG strip on a page is Interpretable. If all 30 minutes of data on the first page are Uninterpretable (noisy or unreadable), the clinician will continue until they find a page of data that includes at least one 30-second strip that is Interpretable. Of the pages that all cardiologists review, a page will be 'Interpretable' if two out of three cardiologists agree that the page is 'Interpretable'; otherwise the page will be 'Uninterpretable' when two out of three agree that the page is 'Uninterpretable'.
Phase 3: Clinical equivalence of ECGs from different electrode placement positions compared to the control position of the Test Device | From enrollment to completion of data collection from all 10 positions performed in a single visit.
  Each subject will undergo 15 minutes of ECG recording under the standard placement (control) and each of the 9 variable placements/Test Positions. The clinical ECG interpretation will be performed by two board-certified cardiologists, with a third involved when there is a disagreement between the two. The cardiologists will provide their assessment for 15-minute recorded data from control and test positions using 'Interpretable' with normal sinus rhythm, ectopy [≤ 3 consecutive beats], or any arrhythmia, or 'Uninterpretable' with noisy or not readable data. Each cardiologist will review the ECGs of subjects from the control and test positions for 'equivalence.' Determination of 'equivalence' will be based on the assessment of the interpretability of the recording. To be equivalent at each 9 test positions, 2 out of 3 cardiologists must agree that the ECGs from control and test positions are 'Interpretable' or 'Uninterpretable.' Otherwise, ECGs are not equivalent.

SECONDARY OUTCOMES:
Test Device Data Quality | Assessments performed after initial application and then 60-minutes and 10-days after application for Phase 1 and Phase 2. For Phase 3, assessments were performed for each of the 10 positions performed in a single day.
  Evaluation of Test Device Data quality graded on a 3-point scale from 0 to 2 categorizing as 0 for good-quality data from all three channels to 2 where channel 2 represents artifacts (not good quality). Tabular summaries of individual subjects' Test Device data quality grades will be summarized for each evaluation time point (All Phases). Descriptive statistics for Test Device data quality grades will be generated for each evaluation time point.
Test Device Skin Adhesion Data | Assessments performed after initial application, 60-minutes after application, and at completion of the 10-day wear time.
  Assessments of skin adhesion of test device adhesive to the skin using a 7-point scale from 0 for being fully adhered to the site to 6 indicating adhesive was completely detached. Tabular summaries of individual subjects' Test Device adhesion grades will be summarized for each evaluation time point (Phase 1 and 2). Descriptive statistics for Test Device adhesion grades will be generated for each evaluation time point.
Skin Condition | Assessments performed after initial application, 60-minutes after application, and at completion of the 10-day wear time
  Visual Evaluations of subjects' skin condition will be assessed using an 8-point scale from 0 representing no evidence of irritation to 7 for strong reactions spreading beyond the test site. Evaluations performed prior to application and 60-minutes after application of the test and reference devices and again after the 10-day wear time of the test device. Tabular summaries of individual subjects' skin condition grades will be summarized for each evaluation (Phase 1 and 2).

OTHER OUTCOMES:
Observations Regarding Test Device Electrode Discoloration / Presence of Particulates | Assessments performed after removal of test day following a 10-day wear time
  For Phase 2 after the 10-wear time, the removed Test Device Adhesives were visually assessed for the presence of any particulates on the side of the adhesive that had been adhered to the subjects' skin. If present, the color and location of particulates were detailed. Tabular summaries of Day 10 (Phase 2) observations regarding Test Device electrode discoloration (including snaps and hydrogel) and the presence of any particulates will be summarized for each individual subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Bioscience of Bozeman, LLC, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans for publishing the data from this trial.